CLINICAL TRIAL: NCT06286579
Title: The Efficacy of New SOI Implant Surface for Immediately Loaded, Post-extractive Versus Delayed Implants
Brief Title: SOI Immediately vs Delayed
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Collaborators: Melodia, Dario, M.D. (Individual); Pisano, Milena, M.D. (Individual); Dr. Aurea M. I. Lumbau (Unknown); Prof. Silvio Mario Meloni (Unknown); Prof. Edoardo Baldoni (Unknown)
Responsible Party: Principal Investigator, Marco Tallarico, Assistant professor, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNISS_PHD_Osstem_3
Record Dates: First submitted 2023-04-24; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Dental Implant; Dental Implant-Abutment Design
Keywords: Dental Implant; Immediately vs Delayes; Implant-abutment connection

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial of parallel group design.
Who Masked: Outcomes Assessor
Masking Description: One "blinded (when possible)" independent assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediately implant placement (Experimental): Atraumatic tooth extraction and immediately placement of implant with a new surface
  Interventions: Device: Immediately implant placement
- Delayed implant placement (Active Comparator): Atraumatic tooth extraction, after the site will be left to heal for 4 months, just grafting with A-Oss and suture, according to a socket preservation procedure. Four month later, implant will be place
  Interventions: Device: Delayed

INTERVENTIONS:
Device: Immediately implant placement — After atraumatic tooth extraction immediate implant placement with SOI surface and loading will be performed with temporary restoration. After osseointegration (8 weeks), the temporary restoration will be modified according to the soft tissue management. After 3 to 4 months, a definitive digital or analog impression will be taken and later definitive restoration will be delivered
  Arms: Immediately implant placement
Device: Delayed — After atraumatic tooth extraction, the extraction site will be left to heal for 4 months, just grafting with A-Oss and suture, according to a socket preservation procedure. Four month later, implant will be place and immediate loadind with temporary restoration will be performed.
  After osseointegration (8 weeks), the temporary restoration will be modified according to the soft tissue management. After 3 to 4 months, a definitive digital or analog impression will be taken and later definitive restoration will be delivered
  Arms: Delayed implant placement

SUMMARY:
The aim of this randomized controlled trial is to compare the clinical and radiographic of immediately loaded, immediate (post-extractive, test group) versus delayed (control group) implants with new SOI surface

ELIGIBILITY:
Inclusion Criteria:

* Any patient with at least one hopeless tooth in the mandible or maxilla, located between premolars, with intact post extractive alveolus. The implants must to engage at least 3 (mandible) to 5 (maxilla) mm of residual native bone over the socket.
* Patients with 18 years or older, and able to sign an informed consent.
* Smokers will be included and categorized into: 1) non smokers; 2) moderate smokers (smoking up to 10 cigarettes/day); 3) heavy smokers (smoking more than 11 cigarettes/day). Heavy smokers will be excluded.
* Biotype will be categorized in thin (≤1 mm), medium (>1 - <2 mm) or thick (≥2 mm).

Exclusion Criteria:

* General contraindications to implant surgery.
* Patients irradiated in the head and neck area.
* Immunosuppressed or immunocompromised patients.
* Patients treated or under treatment with intravenous amino-bisphosphonates.
* Patients with untreated periodontitis.
* Patients with poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Heavy smokers.
* Pregnancy or nursing.
* Substance abuser.
* Psychiatric problems or unrealistic expectations.
* Lack of opposite occluding dentition in the area intended for implant placement.
* Patients with infection and or inflammation in the area intended for implant placement.
* Patients participating in other studies, if the present protocol cannot be properly adhered to.
* Patients referred only for implant placement and cannot be followed ant the treating centre.
* Patients unable to be followed for 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of prosthesis failure | Up to 5 years
  Whether it will not be possible to place the prosthesis because of implant failure or a prosthesis that has to be remade for any reason.
Number of implant failure | Up to 5 years
  defined as implant mobility and/or any infection dictating implant removal, and/or implant fracture and/or any other mechanical complication rendering the implant unusable. The stability of each individual implant will be measured by the local blinded outcome assessors manually tightening the screws with a torque of 30 Ncm at abutment connection, immediately loading, at 1,3 and 5 years after loading for the partial fixed prostheses. Once the single crowns will be cemented, their stability will be assessed by rocking the crown with the handles of two dental instruments.
Number of complications | Up to 5 years
  Technical (fracture of the framework and/or the veneering material, screw loosening, etc.) and/or biologic (pain, swelling, suppuration, peri-implantitis, etc.) complication will be considered.

SECONDARY OUTCOMES:
Rate of peri-implant marginal bone level changes | At 1,3 and 5 years
  Peri-implant marginal bone level changes will be assessed on periapical radiographs took with the paralleling technique at implant placement, at initial loading, 1,3 and 5 years after loading. Ideally digital radiographs should be taken, otherwise radiographs on conventional films will be scanned into TIFF format with a 600 dpi resolution, and stored in a personal computer. Peri-implant marginal bone levels will be measured using the Scion Image (Scion Corporation, Frederick, MD, USA) software. The software will be calibrated for every single image using the known distance of the first two consecutive threads. Measurements of the mesial and distal bone crest level adjacent to each implant will be made to the nearest 0.01 mm. Reference points for the linear measurements will be: the coronal margin of the implant collar and the most coronal point of bone-to-implant contact. Bone levels will be measured.
Valuation of patient satisfaction | At 1,3 and 5 years
  Patients will answer the following questions (separately for each implant):
  1. Are you satisfied with the function of your implant-supported prostheses? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  2. Are you satisfied with the aesthetic outcome of your implant-supported prostheses? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  3. Would you undergo the same therapy again? Possible answers: "yes" or "no".
Rate of implant stability quotient (ISQ) | Up to 5 years
  ISQ was measured and recorded using the IS3 (Osstem), at implant placement, at implants exposure, at the impression time, and prosthetic loading.
Valuation of soft tissue thickness and amount of keratinized tissue | 1,3 and 5 years
  The soft tissue biotype will be investigated by the same surgeon at the surgical procedures using a periodontal probe into the sulcus. Greater will be the thickness of the tissue, smaller will be transparency of the periodontal probe. The amount of keratinized tissue will be evaluated 1 year after surgical procedures using a periodontal probe. This outcome will be evaluated according to the distance from the gingival margin to the mucogingival junction
Number of PES score | 1,3 and 5 years
  Esthetic evaluation of occlusal and vestibular pictures will take every years after definite loading was done following the pink esthetic score (PES). In brief, the PES score evaluates seven variables: mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar process deficiencies, soft tissue color and texture. A 0-1-2 scoring system was used, 0 being the lowest and 2 being the highest value, with a maximum achievable score of 14 per dental unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Tallarico, Sassari, Italy

IPD SHARING:
Plan to Share IPD: No